Official Title: A Comparison of External Ventricular Drain Catheter Diameter on Occlusion and

Replacement: A Randomized Trial

NCT03248739

IRB-Approved Date: 9/12/22



Department/Section of Neurological Surgery

# A COMPARISON OF EXTERNAL VENTRICULAR DRAIN CATHETER DIAMETER ON OCCLUSION AND REPLACEMENT: A RANDOMIZED TRIAL

Informed Consent Form to Participate in Research Kyle M. Fargen, MD, MPH, Principal Investigator

#### Introduction

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you or your loved one has been evaluated by a neurosurgeon and it has been decided that you or your loved one needs an external ventricular drain placed. Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to determine whether the width of an external ventricular drain has any effect on whether it becomes clogged or stops working.

### HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

A total of 120 people at 2 research sites will take part in this study. Approximately 60 will participate at Wake Forest Baptist Health.

#### WHAT IS INVOLVED IN THE STUDY?

Your physician has confirmed that you would benefit from a standard of care catheter called an External ventricular drain (EVD). If you choose to participate in the research study you will be randomized into one of the study groups described below. Randomization means that you are put into a group by chance. It is like flipping a coin. You will have an equal chance of being placed in either group. In the first group, subjects will have a standard of care, FDA approved EVD catheter placed with internal diameter of 1.9mm. In the second group, subjects will have a standard of care, FDA approved EVD catheter placed with internal diameter of 1.5mm. Once you have been randomized into a group, the appropriately sized ventricular catheter will be placed using the standard technique; you will be given medication to help with pain, and the skin of your scalp at the top of your head will be numbed and then cut, a hand-turned drill will be used to drill a hole in your skull, the lining around the brain will be cut, the catheter will be passed at an angle such that it will enter the ventricles in the middle of your brain, and then the end of the catheter outside your head will be tunneled under your scalp and out of the skin



behind the original incision. After placement of the external ventricular drain, a variety of things will be recorded on a daily basis while the catheter is in place, including how often the catheter stops working, how often flushing is required, how often it works, and what the findings are on CT scan if a scan is obtained. The research information collected will be used to determine if the use of one catheter is preferable over the other.

#### How Long WILL I BE IN THE STUDY?

You will be in the study until an attending neurosurgeon decides you no longer need the external ventricular drain.

You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences.

#### WHAT ARE THE RISKS OF THE STUDY?

This study is comparing two different sized approved catheters for treating your condition. You will be randomly assigned to one of the two catheter groups. It is possible that one treatment group may have a better response than the other. Therefore there is a risk that you may be assigned to a group that does not perform as well as its comparison. We don't know at this point which catheter is better. Risks and side effects of this study are the risks and side effects related to your standard of care ventricular catheter placement which include: risk of bleeding, infection, damage to surrounding structures, catheter occlusion, coma, problems with cerebrospinal fluid, paralysis, and transient or permanent loss of all neurological function. You should discuss the risk of being in the study with the study staff.

In addition, there is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. There also may be other side effects that we cannot predict. Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

The Principal Investigator will be responsible for the overall monitoring of the data and safety of study participants. The Principal Investigator will be assisted by other members of the study staff.

## ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

You are not expected to receive any direct benefit from taking part in this research study. We hope the information learned from this study will benefit other people in the future.

#### WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to receive treatment. You should talk to your doctor about all the choices you have. Instead of being in this study, you have the option of allowing your neurosurgeon to choose the catheter and proceed with standard external ventricular drain



management.

WHAT ARE THE COSTS?

All study costs, including any study medications and procedures related directly to the study, will be paid for by the study. Costs for your regular medical care, which are not related to this study, will be your own responsibility.

You or your insurance company will be billed for the standard of care catheter (EVD). You and/or your insurance company will be billed for the cost of any surgical procedure(s) necessary to implant the external drain.

WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified.

Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a research study. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record.

WILL YOU BE PAID FOR PARTICIPATING?

You will receive no payment or other compensation for taking part in this study.

The findings from this research may result in the future development of products that are of commercial value. There are no plans to provide you with financial compensation or for you to share in any profits if this should occur.

WHO IS SPONSORING THIS STUDY?

This study is being sponsored by Wake Forest Department of Neurosurgery.

What Happens if You Experience an Injury or Illness as a Result of Participating in this Study? Should you experience a physical injury or illness as a direct result of your participation in this study, Wake Forest University School of Medicine maintains limited research insurance coverage for the usual and customary medical fees for reasonable and necessary treatment of such injuries or illnesses. To the extent research insurance coverage is available under this policy the reasonable costs of these necessary medical services will be paid, up to a maximum of \$25,000. Wake Forest University Baptist Medical Center holds the insurance policy for this



coverage. It provides a maximum of \$25,000 coverage for each claim and is limited to a total of \$250,000 for all claims in any one year. The Wake Forest University School of Medicine, and the North Carolina Baptist Hospitals, Incorporated do not assume responsibility to pay for these medical services or to provide any other compensation for such injury or illness. Additional information may be obtained from the Medical Center's Director of Risk and Insurance Management, at

If you are injured, the insurer may require information such as your name, social security number, and date of birth in order to pay for your care. This is because the insurer is required by law to report any payments made to cover the care of any persons who are members of a government insurance plan to the Department of Health and Human Services.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Kyle Fargen, MD at

WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any new information we collect from you and/or information we get from your medical records or other facilities about your health or behaviors is considered Protected\_Health Information. The information we will collect for this research study includes: diagnosis, diameter of catheter placed, placement location, level of the EVD, patency, number of times flushed, radiologic outcomes, duration of placement.

If this research study involves the diagnosis or treatment of a medical condition, then Protected Health Information collected from you during this study will be placed in your medical record, and may be used to help treat you, arrange payment for your care, or assist with Medical Center operations.

We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer.

Your personal health information and information that identifies you may be given to others during and after the study. This is for reasons such as to carry out the study, to determine the results of the study, to make sure the study is being done correctly, to provide required reports and to get approval for new products.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board; representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA), the Department of Health and Human Services (DHHS) and similar agencies in other countries.



Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

Monitors, auditors, IRB or other regulatory agencies will be granted direct access to the
participant's original medical record for verification of clinical trial procedures or data,
without violating confidentiality of the participant and to the extent permitted by other
applicable laws.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for an indeterminate period of time. This authorization does not expire. Any research information entered into your medical record will be kept for as long as your medical record is kept by the Medical Center. You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished.

You can tell Kyle Fargen, MD, MPH that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:



However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be



included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information is available to doctors in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Laboratory test results and other medical reports created as a result of your participation in the research study may be entered into the computer systems of Wake Forest University Health Sciences and North Carolina Baptist Hospital. These will be kept secure, with access to this information limited to individuals with proper authority, but who may not be directly involved with this research study.

A North Carolina Baptist Hospital (NCBH) medical record will be created for all study participants. Information about your participation in the study will be placed in the NCBH medical record, along with any routine medical test results that were obtained at NCBH as part of this study.

WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study at any time. This could be because it is in your best medical interest, your condition worsened, new information becomes available, you had an unexpected reaction, you failed to follow instructions, or because the entire study has been stopped.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?
For questions about the study or in the event of a research-related injury, contact the study investigator, Kyle Fargen, MD at \_\_\_\_\_\_\_.

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at



You will be given a copy of this signed consent form.

#### **S**IGNATURES

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| Subject Name (Printed): | <del></del> | | |
|---|---|---|---|
| Subject Signature: | Date: | Time: | am pm |
| Person Obtaining Consent (Printed): | | | |
| Person Obtaining Consent: | Date: | Time: | am pm |
| Legally Authorized Representative Name (Pri | nt): | | |
| The above named Legally Authorized Represe subject based upon (specify health care power | _ | • | e research |
| Relationship to the Subject: | | | |
| Legal Representative Signature: | Date: | Time: | am pm |